CLINICAL TRIAL: NCT05830630
Title: The Preventive Value of Continuous Perineural Methylene Blue Infusion in Patients Undergoing Lower Limb Amputation Surgery
Brief Title: Perineural Methylene Blue Infusion in Lower Limb Amputation Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, lecturer of anesthesiology, surgical intensive care and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264PR174/4/23
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Perineural; Methylene Blue; Lower Limb Amputation
Keywords: Perineural; Methylene blue; Lower limb amputation

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine methylene blue group (Experimental): Patients in this group will receive the following regimen through the perineural catheter:
  Bolus dose of 1 ml methylene blue 1% (10 mg) plus 19 ml bupivacaine 0.25% will be given intraoperatively before wound closure, and perineural infusion of methylene blue plus bupivacaine 0.25% (1 ml of methylene blue added to each 49 ml of bupivacaine 0.25%) will be started in the recovery room at a rate of 2-5 ml/hour for 72 hours postoperatively
  Interventions: Drug: Bupivacaine methylene blue
- Bupivacaine saline group (Active Comparator): Patients in this group will receive the following regimen through the perineural catheter:
  Bolus dose of 1 ml normal saline plus 19 ml bupivacaine 0.25% will be given intraoperatively before wound closure, and perineural infusion of bupivacaine 0.25% will be started in the recovery room at a rate of 2-5 ml/hour for 72 hours postoperatively
  Interventions: Drug: bupivacaine saline

INTERVENTIONS:
Drug: Bupivacaine methylene blue — Patients in this group will receive the following regimen through the perineural catheter:
  Bolus dose of 1 ml methylene blue 1% (10 mg) plus 19 ml bupivacaine 0.25% will be given intraoperatively before wound closure, and perineural infusion of methylene blue plus bupivacaine 0.25% (1 ml of methylene blue added to each 49 ml of bupivacaine 0.25%) will be started in the recovery room at a rate of 2-5 ml/hour for 72 hours postoperatively
  Arms: Bupivacaine methylene blue group
Drug: bupivacaine saline — Patients in this group will receive the following regimen through the perineural catheter:
  Bolus dose of 1 ml normal saline plus 19 ml bupivacaine 0.25% will be given intraoperatively before wound closure, and perineural infusion of bupivacaine 0.25% will be started in the recovery room at a rate of 2-5 ml/hour for 72 hours postoperatively
  Arms: Bupivacaine saline group

SUMMARY:
This prospective randomized controlled study will be conducted to evaluate the analgesic effect of continuous perineural infusion of methylene blue with bupivacaine on acute postoperative pain and to evaluate its preventive role against chronic phantom pain in patients undergoing lower limb amputation surgery

DETAILED DESCRIPTION:
Post amputation pain remains an extremely challenging pain condition to treat, so the prevention of phantom pain is our goal to decrease its incidence.

Methylene blue, an inhibitor of nitric oxide synthase and guanylate cyclase, has been widely applied for a variety of pain-related diseases due to its characteristic abilities, such as the blocking of pain transmission, antioxidant, and anti-inflammatory effects. Methylene blue can maintain local anesthesia for approximately 20 days so it can be used as a nerve block to relieve pain, especially refractory neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, suffering from vascular insufficiency of one or both lower limbs and scheduled for above or below knee amputation under general anesthesia.

Exclusion Criteria:

* Patients with a history of allergy to local anesthetics.
* Patients with allergy to methylene blue.
* Anticoagulant use or coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Degree of postoperative pain | 3 days after surgery
  Degree of postoperative pain will be assessed using visual analogue scale which is a 10 cm scale ranging from (0 = no pain to 10 = worst possible pain)

SECONDARY OUTCOMES:
Incidence of phantom limb pain | 9 months after surgery
  Incidence of phantom limb pain at day 6 after surgery then at 1, 3, 6, 9 months after surgery

OTHER OUTCOMES:
Incidence of stump pain | 9 months after surgery
  Incidence of stump pain at day 6 after surgery then at 1, 3, 6, 9 months after surgery
Postoperative opioid consumption | 3 days after surgery
  Morphine consumption in the 1st 3 days after surgery will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available upon a reasonable request from the corresponding author after the end of study for 1 year
Access Criteria: The data will be available upon a reasonable request from the corresponding author